CLINICAL TRIAL: NCT05209412
Title: Paclitaxel-Coated Balloon Versus Zotarolimus-Eluting Stent for Treatment of De Novo Coronary Artery Lesions: an Open-label, Multicenter, Randomized, Non-inferiority Trial
Brief Title: Paclitaxel-Coated Balloon Versus Zotarolimus-Eluting Stent for Treatment of De Novo Coronary Artery Lesions
Acronym: CAGE-FREEIII
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, LingTao, Professor in Cardiology, Director of the department of Cardiology, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAGE-FREE III
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: De Novo Stenosis; Coronary Artery Disease; Percutaneous Coronary Intervention
Keywords: Drug-coated balloons; Fractional flow reserve; Percutaneous coronary intervention; De novo lesions; Drug-eluting stent
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin; Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug-coated balloon (Experimental): Lepu Paclitaxel coated balloon will be used
  Interventions: Device: Lepu Paclitaxel coated balloon; Drug: Aspirin; Drug: Ticagrelor; Drug: Clopidogrel
- Drug-eluting stent (Active Comparator): Resolute Integrity Zotarolimus eluting stents will be used
  Interventions: Device: Resolute Integrity Zotarolimus eluting stents; Drug: Aspirin; Drug: Ticagrelor; Drug: Clopidogrel

INTERVENTIONS:
Device: Lepu Paclitaxel coated balloon — Paclitaxel is the pharmacologically active substance for anti-neointima. The active drug coating is located on the surface of the balloon, which contains 1.5 μg Paclitaxel per 1 mm2.
  Arms: Drug-coated balloon
Device: Resolute Integrity Zotarolimus eluting stents — The device consists of a balloon-expandable intracoronary drug-eluting stent pre-mounted on the MicroTrac Rapid Exchange stent delivery system. Drug eluting stent is composed of metal stent, primer and drug coating. The Stent is manufactured from a cobalt alloy (MP35N). The strut thickness is 88.9 μm and the length elements is 0.9 mm. The drug coating consists of the zotarolimus and BioLinx polymer (C10/C19/PVP) system. A coating of polymers loaded with zotarolimus in a formulation applied to the entire surface of the stent at a dose of approximately 1.6 µg/mm2 which results in a maximum nominal drug content of 380 µg on the largest stent (4.0 x 38 mm).
  Arms: Drug-eluting stent
Drug: Aspirin — Aspirin is required for 3 months be a part of the dual antiplatelet therapy (DAPT) after PCI.
Drug: Ticagrelor — Ticagrelor is required for 12 months to be a part of the dual antiplatelet therapy (DAPT) after PCI.
Drug: Clopidogrel — Clopidogrel is required for 12 months to be a part of the dual antiplatelet therapy (DAPT) after PCI when Ticagrelor is unfeasible or contradicted.

SUMMARY:
Coronary restenosis has been one of the main reasons affecting the prognosis of patients with coronary artery disease (CAD) after percutaneous coronary intervention (PCI). With drug-eluting stents (DES), which elutes an antiproliferative drug to the vessel wall and reduces the restenosis rate; however, the incidence of restenosis is still about 10%. The late stent thrombosis and restenosis, with a hazard of nearly 2% per year after implantation, remained a concern and motivated the development of drug-coated balloons (DCB).

DCB angioplasty has the following advantages compared with DES implantation: Firstly, the drug in DCB is uniformly distributed and released; whereas the drug release of DES via stent platform is uneven -85% of the vascular wall is not covered by the stent strut. Secondly, there is no alloy in the vessel after DCB angioplasty, while the coronary stent platform and polymer might cause temporal or persistent inflammatory response leading to intimal hyperplasia. Finally, there is no metal cage restraining vessel motion after DCB, the physiological function of coronary arteries would be maintained.

Studies with the strategy of DCB angioplasty with bailout stenting have demonstrated safety and efficacy for the small-vessel disease. The application of DCB in large vessels with de novo lesions is still to be investigated. The DEBUT study showed that in high bleeding risk patients aimed using only 1-month DAPT, DCB was superior to BMS in terms of MACE [MACE (cardiovascular mortality, nonfatal myocardial infarction or revascularization of ischemia-reperfusion target lesions)] at 9-month follow-up.

However, there is still a lack of evidence comparing the DCB versus DES in large vessels with de novo lesions. The current study aims to investigate if in patients undergoing PCI for de novo stenoses in large vessels, DCB is non-inferior to DES.

ELIGIBILITY:
Inclusion Criteria:

1. 18y ≤ age ≤ 80y;
2. De-novo coronary artery lesions with an indication for PCI;
3. Target lesion diameter stenosis ≥ 70% (visual) or ≥ 50% (visual) with evidence of ischemia;
4. Target lesion reference vessel diameter (2.5mm-4.0 mm), Length of a single target lesion ≤ 35mm; Total treated lesion length ≤ 60 mm;
5. Vessels treated ≤ 2; only one DCB/DES is allowed for each target vessel;
6. ≤ 2 non-target lesions (non-TL) are allowed, and can not be in the same vessel as the target lesion (randomization should be implemented only after the successful treatment of all non-TL);
7. Patients who are able to complete the follow-up and compliant to the prescribed medication.

Exclusion Criteria:

1. Myocardial infarction (< 7 days);
2. Heavy thrombotic burden in target vessel;
3. eGFR < 30ml/min or hemodialysis patients;
4. Other cardiovascular and cerebrovascular procedures planned within 12 months after index PCI;
5. Patients with contraindications to antiplatelet agents and anticoagulants or bleeding tendency, history of active peptic ulcer, and stroke within 6 months;
6. Life expectancy of less than 1 years;
7. Patient is a woman who is pregnant or nursing;
8. Known allergic to medications such as Aspirin, Heparin, antiplatelet drugs, paclitaxel, or contrast; patients with systemic lupus erythematosus or other systemic immune diseases;
9. Chronic total occlusion lesion;
10. Unprotected left main disease;
11. Bifurcation lesion requiring 2 stents;
12. Ostial lesions, distance from left main ≤ 2mm;
13. Severe calcification or distortion;
14. Arterial, venous or prosthetic grafts;
15. In-stent stenosis requiring revascularization (defined as stenosis≥50% by visual or positive functional assessments in any vessel);
16. Myocardial bridging located at target lesions;
17. Currently participating in another trial and not yet at its primary endpoint;
18. Participants deemed unsuitable to be enrolled by investigators for unable to comply with protocol or other reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Coronary fraction flow reserve (FFR) value | 12 months

SECONDARY OUTCOMES:
In segment Late lumen loss (LLL) | 12 months
  Key Secondary Outcome

OTHER OUTCOMES:
Procedural success rate | 7 days
  Procedural success rate included device success, lesion success and procedural success
Percentage of lesion segments diameter stenosis (DS%) | 12 months
Binary restenosis (DS% ≥ 50%) | 12 months
Target lesion failure (TLF) | 1, 6, 12 months
  Target lesion failure (TLF), defined as cardiac death, target vessel myocardial infarction (TV-MI) and clinically indicated-target lesion revascularization (CI-TLR)
Patient-oriented composite endpoint (PoCE) | 1, 6, 12 months
  Patient-oriented composite endpoint (PoCE) defined as all-cause death, any stroke, any MI, and any clinically and indicated revascularisation)
Definite/Probable Stent thrombosis rates | 1, 6, 12 months
  Stent thrombosis included acute, subacute, late and very late thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, M.D, Ph.D, Study Chair — Xijing Hospital; Chao Gao, M.D, Ph.D, Study Chair — Xijing Hospital
Locations (1):
- Ling Tao, Xi'an, Shannxi, China